CLINICAL TRIAL: NCT04938193
Title: 68Gallium-citrate Positron Emission Tomography/Computed Tomography (68Ga-citrate PET/CT) for the Diagnosis of Chronic Prosthetic Hip or Knee Infection
Brief Title: 68Ga-citrate PET/CT for the Diagnosis of Chronic Prosthetic Hip or Knee Infection
Acronym: Gal-I-TEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/24
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-citrate PET/CT (Experimental)
  Interventions: Diagnostic Test: 68Ga-citrate PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-citrate PET/CT — PET/CT Imaging with 68Ga-citrate PET/CT injection

SUMMARY:
Diagnosis of chronic prosthetic joint infection (PJI) can be difficult. 68Ga-citrate Positron Emission Tomography/Computed Tomography (PET/CT) has been recently developed and has many advantages such as high resolution and low radiation exposure. To date, 68Ga-citrate PET/CT has not been specifically assessed in prosthetic joint infection. In this prospective study, patients referred for a suspected PJI will benefit from both a 68Ga-citrate PET/CT and a 99mTc-HMPAO-labelled leukocyte SPECT/CT. The primary outcome is the assessment of the 68Ga-citrate PET/CT accuracy for the diagnosis of chronic prosthetic hip or knee infection.

DETAILED DESCRIPTION:
Prosthetic joint infection (PJI) is a serious and rare complication of orthopedic surgery. Diagnosis is based on precise criteria (MSIS criteria Musculoskeletal Infection Society). However, diagnosis can be difficult, in particular when the infection is present for more than one month. One of the usual exams is bone scintigraphy and 99mTc-HMPAO-labelled leukocyte scintigraphy. This imaging allows an accurate assessment but it has some limitations since it requires ex vivo isolation and marking of patient's leukocytes and repeated acquisition for 24 hours. 68Gallium-citrate positron emission tomography/computed tomography (68Ga-citrate PET/CT) has been recently developed. 68Ga-citrate PET/CT is innovative compared to [18F]fluorodeoxyglucose PET/CT (18F-FDG PET/CT) and has many advantages: high resolution, realization in only two hours, short radioactive period and no handling of patient's leukocytes. Furthermore, preliminary data indicate that 68Ga-citrate is picked up by immune cells, which makes this exam inflammation-selective. To date, 68Ga-citrate PET/CT has not been specifically assessed in PJI, it is the objective of the present study:

Prospective study using 68Ga- citrate PET/CT and a 99mTc-HMPAO-labelled leukocyte SPECT/CT. Patients referred for a suspected PJI and with a positive bone scintigraphy will be prospectively enrolled. After information and signature of informed consent, patients will benefit from a 68Ga citrate PET/CT, in addition to leukocyte scintigraphy in a two-week period. Both images will be anonymized and interpreted by two independent nuclear physicians.

Final PJI diagnosis is based on reference criteria (MSIS) to ensure diagnosis during the standardized medical follow-up. Patients will be followed until 12 months after the leukocyte scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Patient referred for the first time to the South-Western France referral center for complex bone and joint infections (Crioac GSO, infectious diseases and orthopedic surgery units) for suspicion of prosthetic hip or knee infection.
* Suspicion of prosthetic joint infection evolving for more than one month.
* Patient for who routine diagnosis includes both bone scintigraphy and leukocytes scintigraphy.
* Patient with positive bone scintigraphy.
* Being affiliated to a health insurance system
* Having signed an informed consent form (later than the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Patient with active cancer.
* Patient with negative bone scintigraphy.
* Patient who cannot stop antibiotics 14 days before exams.
* Pregnant or breastfeeding women.
* Women of childbearing age but not using effective means of contraception.
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).
* Subject in relative exclusion period from another study protocol.
* Known contraindications to PET exam with radiopharmaceutical injection (hypersensitivity to radiopharmaceutical and/or to excipients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 68Ga citrate PET / CT scan CT for chronic prosthetic hip or knee infection | Up to 12 months after baseline (Day 0)
  Sensibility, specificity, positive and negative predictive value. Index test : 68Ga citrate PET / CT scan CT at inclusion. Reference test : Musculoskeletal Infection Society (MSIS) criteria assessed up to 12 months after inclusion. After 12 months, participants will be considered free of chronic prosthetic hip or knee infection.

SECONDARY OUTCOMES:
Diagnostic accuracy of quantitative 68Ga citrate PET / CT scan for chronic prosthetic hip or knee infection | Up to 12 months after baseline (Day 0)
  Area under ROC curve (AUROC) for SUVmax ROI and SUVmax ROI/SVmax liver region ratio measured at inclusion.
  Reference test : Musculoskeletal Infection Society (MSIS) criteria assessed up to 12 months after inclusion.
Inter-observer reproducibility of 68Ga-citrate PET/CT interpretation | Up to 12 months after baseline (Day 0)
  Intraclass correlation coefficient and/or Cohen's Kappa.
Diagnostic accuracy of leukocyte scintigraphy for chronic prosthetic hip or knee infection | Up to 12 months after baseline (Day 0)
  Sensibility, specificity, positive and negative predictive values. Index test : leukocytes scintigraphy at inclusion. Reference test : Musculoskeletal Infection Society (MSIS) criteria assessed up to 12 months after inclusion.
Diagnosis accuracy of 68Ga-citrate PET/CT and leukocytes scintigraphy for chronic prosthetic hip or knee infection in the following sub-groups: prosthetic knee or hip infection. | Up to 12 months after baseline (Day 0)
  Sensibility, specificity, positive and negative predictive values, in each subgroup.
  Index test : 68Ga citrate PET / CT scan CT at inclusion. Reference test : Musculoskeletal Infection Society (MSIS) criteria assessed up to 12 months after inclusion. After 12 months, participants will be considered free of chronic prosthetic hip or knee infection.
Comparison of diagnostic accuracy of 68Ga-PET/CT and leukocytes scintigraphy for chronic prosthetic hip or knee infection | Up to 12 months after baseline (Day 0)
  Sensibility, specificity, positive and negative predictive values. Reference test : Musculoskeletal Infection Society (MSIS) criteria assessed up to 12 months after inclusion.
  Index test : 68Ga citrate PET / CT scan CT at inclusion and leukocytes scintigraphy at inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric-Antoine DAUCHY, MD, Principal Investigator — University Hospital, Bordeaux; Eric FRISON, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de maladies infectieuses, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No